CLINICAL TRIAL: NCT00703872
Title: An Evaluation of Two Dose Routes of HDV-Interferon Administered With Ribavarin in the Treatment of Chronic Hepatitis C Nonresponders and Naive Hepatitis C Patients
Brief Title: HDV-Interferon in the Treatment of Chronic Hepatitis C Nonresponders and Naive Hepatitis C Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hepasome Pharmaceuticals (Industry)
Responsible Party: Len Rosenberg, PhD, RPh, Hepasome Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP 01-2006-01
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Naive; Nonresponders; Interferon; Patients with Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral HDV-Interferon
  Interventions: Drug: Oral HDV-Interferon + ribavarin
- 2 (Experimental): Injectable HDV-Interferon + ribavarin
  Interventions: Drug: Injectable HDV-Interferon + ribavarin

INTERVENTIONS:
Drug: Oral HDV-Interferon + ribavarin — Naive pateints
  Arms: 1
Drug: Injectable HDV-Interferon + ribavarin — Nonresponders
  Arms: 2

SUMMARY:
A Phase II, Open Label, Multi-Center, Proof-Of-Concept Study determing whether treatment with HDV-Interferon (HDV-IFN), by oral or subcutaneous (injection) routes, and ribavirin results in similar efficacy [Rapid Virologic Response (RVR)] and safety as the reported efficacy and safety with pegylated alpha-interferon-2a and ribavirin (historical control) in patients with chronic hepatitis C (treatment naïve by oral route and non-responders by SC route respectively).

DETAILED DESCRIPTION:
Part 1 ("initial part") - 4 weeks of treatment (28 days):

* All patients will complete an initial 4 weeks of treatment with HDV-Interferon (HDV-IFN) (treatment naïve by oral route and non-responders by SC route respectively) and ribavirin.
* The Part 1 of the study shall assess whether a 4-week treatment course with HDV-Interferon (HDV-IFN), orally or by subcutaneous injection, and ribavirin results similar efficacy [Rapid Virologic Response (RVR)] and safety as the reported efficacy and safety with pegylated alpha-interferon-2a and ribavirin (historical control) in patients with chronic hepatitis C (treatment naïve and non-responders).

Part 2 ("continuation part") - 44 or 20 weeks of treatment + 24 weeks (follow-up period):

* Patients with hepatitis C viral genotype 1, who achieve RVR, will be treated for another 44 weeks of therapy (to complete 48 weeks of active treatment) followed by 24 weeks of treatment-free follow-up period.
* Patients with hepatitis C viral genotype 3, who achieve RVR, will be treated for another 20 weeks of therapy (to complete 24 weeks of active treatment) followed by 24 weeks of treatment-free follow-up period.
* Follow-up period (24 weeks): Thus, in addition to treatment in Part 1 of study, each completed patient with viral genotype 1 will receive 44 weeks of therapy and 24 weeks of treatment-free follow-up; and viral genotype 3 patients will have 20 weeks of therapy & 24 weeks of treatment study drug free follow-up.
* Overall study duration (72 or 48 weeks): Patients with viral genotype 1 will have an overall study duration of 72 weeks (48 weeks of therapy plus 24 weeks follow-up) and patients with viral genotype 3 will have an overall study duration of 48 weeks (24 weeks of therapy plus 24 weeks follow-up).

ELIGIBILITY:
Inclusion Criteria - Nonresponders:

* Patients >18 years with established chronic hepatitis C with viral genotype 1 or viral genotype 3 who have failed to respond to at least a 3-month course of a pegylated interferon alpha 2a + ribavirin and have a detectable HCV RNA and baseline liver biopsy available from within the prior 12 months.

Inclusion Criteria - Naive:

* Treatment naïve patients > 18 years, inclusive, are eligible for this study.
* Patients will be viral genotype 1 or viral genotype 3, have quantifiable HCV-RNA > 1000 IU/mL as demonstrated by PCR and an abnormal ALT (within 6 months of screening) and compensated liver disease with or without cirrhosis.

Exclusion Criteria - Nonresponders:

* Patients with decompensated cirrhosis or other forms of liver disease
* Hb < 10g/dL for males & Hb < 9 g/dl for females
* hepatocellular carcinoma
* active hepatitis B infection
* human immunodeficiency virus (HIV)
* pre-existing severe or uncontrolled depression or other psychiatric disease
* significant cardiac disease
* renal disease
* seizure disorders or retinopathy

Exclusion Criteria - Nonresponders:

* Patients with decompensated cirrhosis or other forms of liver disease
* Hb < 10g/dL for males & Hb < 9 g/dl for females
* hepatocellular carcinoma
* active hepatitis B infection
* HIV
* pre-existing severe or uncontrolled depression or other psychiatric disease - significant cardiac disease
* renal disease
* seizure disorders or retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Rapid Virologic Response | 4 weeks

SECONDARY OUTCOMES:
Early Virologic Response | 12 Weeks
Sustained Virologic Response | 24 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dharmesh Kapoor, MD, Principal Investigator — Global Hospitals, Lakdi-ka-pool, Hyderabad - 500 004 India
Locations (1):
- Global Hospitals, Lakdi-ka-Pool, Hyderabad, India